CLINICAL TRIAL: NCT07072299
Title: DEB-BACE for Primary Lung Cancer: A Retrospective, Single-Arm, Multicenter Study on Efficacy and Safety
Status: Not yet recruiting | Type: Observational
Sponsor: Gang Wu, MD (Other)
Responsible Party: Sponsor-Investigator, Gang Wu, MD, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Other Study IDs: 2025-KY-0872-001
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Lung Cancer Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: DEB-BACE — Drug-Eluting Bead microspheres used for embolization: Drug-Eluting Bead microspheres 1tube was loaded and adsorbed chemotherapy. End point of embolization: stagnation of blood flow in tumor feeding artery

SUMMARY:
This is a retrospective, single-arm, multicenter clinical study designed to evaluate the efficacy and safety of DEB-BACE (Drug-Eluting Bead Bronchial Artery Chemoembolization) in the treatment of primary lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old, gender unrestricted; 2. Diagnosed with primary lung cancer based on the Primary Lung Cancer Diagnosis and Treatment Guidelines (2022 Edition) through histopathological examination; 3. At least one measurable lesion (evaluated according to RECIST 1.1 criteria); 4. Previously received at least one DEB-BACE treatment; 5. ECOG PS score ≤ 2; 6. Complete patient case records.

Exclusion Criteria:

* 1. Presence of extensive and uncontrolled extrapulmonary brain metastasis lesions; 2. Irreversible coagulation dysfunction within a short period of time; 3. Uncontrollable hypertension, diabetes, or significant cardiovascular diseases with obvious symptoms; 4. Allergy to contrast agent; 5. Pregnant or lactating women; 6. Patients whose condition, as judged by the investigator, poses a serious threat to patient safety or hinders their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Lung Cancer
Sampling Method: Non-Probability Sample
Enrollment: 1213 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 1 years
  ORR is defined as the percentages of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to mRECIST 1.1 criteria

SECONDARY OUTCOMES:
PFS | up to 1 years
  PFS was defined as the time from recruitment to the first documented progressive disease (PD) or death due to any cause, whichever occurred first.
OS | up to1 years
  The time from recruitment to death due to any cause

IPD SHARING:
Plan to Share IPD: No